CLINICAL TRIAL: NCT03939416
Title: Study of the Influence of Manual Therapy According to the POLD Method Within a Pain Treatment Program in Fibromyalgia
Brief Title: Study of the Influence of POLD Manual Therapy in Fibromyalgia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participants were recruited for a quality study
Sponsor: Omphis Foundation (Other)
Collaborators: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Juan Vicente, López Díaz, Director, Omphis Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pold-fibromyalgia-udl
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Chronic pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POLD concept treatment (Experimental): Patients treated with rhythmic mobilizations according to the POLD concept, in addition to the standart treatment
  Interventions: Other: Experimental
- CONTROL (Active Comparator): Patients treated with the standart treatment
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — STANDART
  1. Physical exercise: degreed joint mobilization, self muscle elongation and postural correction.
  2. Sophrology: mental control of insomnia and painful perception
  3. Cognitive behavioral therapy: analysis of non-assertive relationship patterns or dependence, dysfunctional beliefs, as well as their consequences, psychoeducation of the disease. Strategies for pain management, anxiety, assertiveness and acceptance of the disease
  POLD
  1. Rhythmic transversal muscle mobilization in posterior chain musculature.
  2. General vertebral decompression from the sacrum and pelvis
  3. Metameric subcutaneous mobilization
  4. Rhythmic vertebral mobilization from the spinous processes.
  Other Names: POLD concept treatment + standart treatment
  Arms: POLD concept treatment
Other: Control — STANDART
  1. Physical exercise: degreed joint mobilization, self muscle elongation and postural correction.
  2. Sophrology: mental control of insomnia and painful perception
  3. Cognitive behavioral therapy: analysis of non-assertive relationship patterns or dependence, dysfunctional beliefs, as well as their consequences, psychoeducation of the disease. Strategies for pain management, anxiety, assertiveness and acceptance of the disease
  Other Names: Standart treatment
  Arms: CONTROL

SUMMARY:
This clinical research aims to study the effects of the introduction of POLD manual therapy within the protocol of fibromyalgia

DETAILED DESCRIPTION:
This research project aims to generate scientific evidence on the clinical results obtained in the treatment of fibromyalgia, which usually presents with pain and long-term disability, by applying a special form of manual physiotherapy called "POLD concept". This therapy is based on a passive, oscillatory mobilization, performed at a resonance frequency and applied throughout the time of the therapeutic session, on the vertebrae and the muscles of the back, without interruption. It is carried out on the initiative of the research team in "pain treatment", of the physiotherapy school of the University of Lleida, in collaboration with the Omphis Foundation and the clinical service of the Unity of Fibromyalgia of GSS (Hospital Universitarios de Santa María, Lleida)

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Fibromyalgia
2. Patients over 25 years old and up to 65 years old, regardless of whether they are women or men.
3. Patients who present pain with a minimum value of 5 on the numerical pain scale from 0 to 10, at the time of beginning the study.
4. Presence of these symptoms in a long period (more than 6 months)

Exclusion Criteria:

1. Patients with a recent traumatic history.
2. Presence of an irradiation component of neurological origin to upper or lower limbs
3. Patients with neurological alterations, both central and peripheral.
4. Patients who are taking opioid-based analgesic medication.
5. Patients with severe spinal malformations.
6. That they are following any other type of treatment, whether manual or physical agents or alternative or complementary therapies.
7. That they have been treated with infiltrations or similar in a period of less than one year before beginning the study.
8. Patients with a serious psychiatric history such as schizophrenia or psychopathies.
9. Patients who have vestibular problems that do not tolerate oscillation.
10. Patients with heart failure
11. Existence of judicial process of disability

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Demographic data | Participants will be followed for the duration of treatment application, an expected average of 8 weeks.
  The following data will be recorded: age, sex, race, children, study start date and final date.
Level of Pain: VAS | Participants will be followed for the duration of treatment application, an expected average of 8 weeks.
  We will use the Visual Analog Pain Scale (VAS), consisting of a line of 10 cm, whose left end coincides with the value 0 (absence of pain) and the right end with the value 10 (maximum pain imaginable), without reference marks intemediate The patient will mark a point in the line corresponding to his pain at the time of the test, the measurement of the centimeters from the left edge will indicate the analogical score of his pain between 0 and 10.
Quality of pain: The Mc Gill pain questionnaire | Participants will be followed for the duration of treatment application, an expected average of 8 weeks.
  The Mc Gill pain questionnaire comprises 62 descriptors distributed in 15 classes and, in turn, in 3 dimensions (sensory, affective and evaluative).
  A value of pain is obtained for each dimension: sensory pain intensity (VID (S), affective pain intensity (VID (A)) and evaluative pain intensity (VID (E)) The sensory component is evaluated in 7 subclasses. The patient mark one or no descriptor of each subclass, if he scores 1 he scores 1 and if he does not mark none he scores 0. The score of the VID (S) is obtained adding and will be, therefore, between 0 and 7. The affective dimension includes subclasses 8 to 13 and its score ranges from 0 to 6. The evaluative dimension corresponds to subclass 14 and the score of it will be 0 or 1. From the sum of the three, the total score (VID (T)) is obtained, from 0 to 14. In addition, the current pain intensity (VIA) is scored from subclass 15, the score is 0-no pain, 1-mild, 2-annoying, 3-intense, 4-strong, 5-unbearable.
Pain interference: We use the Brief Pain Inventory | Participants will be followed for the duration of treatment application, an expected average of 8 weeks.
  We use the Brief Pain Inventory that gives two main scores: a pain severity score and a pain interference score. The pain severity score is calculated from the four items about pain intensity. Each item is rated from 0, no pain, to 10, pain as bad as you can imagine, and contributes with the same weight to the final score, ranging from 0 to 40. The pain interference score corresponds to the item on pain interference. The seven sub items are rated from 0, does not interfere, to 10, completely interferes, and contributes with the same weight to the final score, ranging from 0 to 70. The first item, pain drawing diagrams (painful and most painful areas) do not contribute to the scoring

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Campoy, PHD, Principal Investigator — Universitat se Lleida; Juan Vicente López Díaz, PHD, Study Director — Universitat de Lleida
Locations (1):
- Specialized hospital unit of fibromyalgia and SD of conical fatigue of L'Hospital Universitari de Santa María (GSS), Lleida, Catalonia, Spain